CLINICAL TRIAL: NCT01194284
Title: Observational, Noninterventional Surveillance Study of Patients With Newly Diagnosed Osteosarcoma
Brief Title: Surveillance Study of Patients With Newly Diagnosed Osteosarcoma
Status: Terminated | Type: Observational
Why Stopped: Regulatory agency commitment fulfilled.
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: C23003; 2009-017204-89 (EudraCT Number)
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — mifamurtide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- High-grade osteosarcoma patients
  Interventions: Drug: Mifamurtide

INTERVENTIONS:
Drug: Mifamurtide — Mifamurtide will be prescribed to patients with high-grade osteosarcoma as part of their treatment regimen within the context of prevailing standard oncology practice. The recommended dose of mifamurtide is 2 mg/m2. Mifamurtide will be administered for 36 weeks as adjuvant therapy following surgical resection.
  Other Names: MEPACT

SUMMARY:
This study is an observational safety surveillance study designed to prospectively assess patients with high-grade osteosarcoma who are candidates for treatment with mifamurtide within the context of prevailing standard oncology practice

ELIGIBILITY:
Inclusion Criteria

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Male or female aged 2 to 40 years
* Confirmed pathological diagnosis of newly-diagnosed, nonmetastatic, resectable, primary, high-grade osteosarcoma
* Have completed definitive surgery (or other local ablation technique)
* Have a treatment regimen that includes mifamurtide and a minimum of 2 recognized chemotherapy agents in the treatment of osteosarcoma (cisplatin, doxorubicin, high-dose methotrexate or ifosfamide)
* Organ function deemed satisfactory to receive planned chemotherapy containing at minimum 2 of the recognized chemotherapy agents in the treatment of osteosarcoma
* Voluntary Written Consent

Exclusion Criteria

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Female patients who are lactating and breastfeeding or have a positive serum pregnancy test during the screening period
* History of pericarditis or pleuritis
* Have low-grade osteosarcoma or parosteal or periosteal sarcoma
* Have osteosarcoma associated with Paget's disease
* Current treatment with any anticancer investigational products at the time of enrollment in this study

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of patients with high-grade osteosarcoma who are candidates for treatment with mifamurtide within the context of prevailing standard oncology practice.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Short-term safety profile of mifamurtide during treatment (mifamurtide in combination with chemotherapy) | 36 weeks
  * Adverse events of special interest (AESIs), including important identified and potential risks
  * The frequency and pattern of mifamurtide-related infusion adverse events
The long-term safety profile of mifamurtide during and following treatment (mifamurtide in combination with chemotherapy) | Up to 5 years from the last dose of mifamurtide or until death
  Assessment of AESIs, consisting of important identified and potential risks

SECONDARY OUTCOMES:
Disease-free survival | Up to 5 years from the last dose of mifamurtide or until death
Overall Survival | Up to 5 years from the last dose of mifamurtide or until death

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- AKH Wien Universitätsklinik für Innere Medizin I Klinische Abteilung für Onkologie, Vienna, Austria